CLINICAL TRIAL: NCT02399267
Title: The Frequency of Screening and SBT Technique Trial
Brief Title: Frequency of Screening and SBT Technique Trial
Acronym: FAST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Screening
Other Study IDs: FAST-001
Record Dates: First submitted 2015-03-15; First posted 2015-03-26 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Critically Ill
Keywords: mechanical ventilation; weaning; critically ill; spontaneous breathing trial; screening; invasive ventilation; SBT technique
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Once daily screening (Active Comparator): In the 'once daily screening arm', RTs will screen invasively ventilated patients between approximately 06:00 - 08:00 hours daily. If a screening period is missed inadvertently or due to an investigation or intervention (operation/procedure) necessitating absence from the ICU, it may be conducted later on the same day and ideally within 6 hours of the scheduled screening period. Regardless of group assignment, if the SBT screening assessment is passed, an SBT will be conducted as per protocol.
  Interventions: Procedure: Once daily screening
- At least twice daily screening (Experimental): In the 'at least twice daily' screening arm patients will be screened at a minimum between approximately 06:00 - 08:00 hours and 13:00 - 15:00 hours daily. If a screening period is missed inadvertently or due to an investigation or intervention (operation/procedure) necessitating absence from the ICU, it may be conducted later on the same day and ideally within 6 hours of the scheduled screening period. Additional screening trials in the 'at least twice daily' screening arm will be permitted at the discretion of the clinical team (RTs and physicians). Regardless of group assignment, if the SBT screening assessment is passed, an SBT will be conducted as per protocol.
  Interventions: Procedure: Twice daily screening
- PS SBTs (Active Comparator): In the 'PS SBTs arm', RTs will conduct SBTs using only PS =< 8 cm H2O with PEEP =< 5 cm H2O. Regardless of group assignment, if the SBT screening assessment is passed, an SBT will be conducted as per protocol.
  Interventions: Procedure: PS SBTs
- T-piece SBTs (Active Comparator): In the 'T-piece SBTs arm', RTs will conduct SBTs using only T-piece. Regardless of group assignment, if the SBT screening assessment is passed, an SBT will be conducted as per protocol.
  Interventions: Procedure: T-piece SBTs

INTERVENTIONS:
Procedure: Once daily screening — RTs will screen invasively ventilated patients between approximately 06:00 - 08:00 hours daily. To pass the 'readiness to wean screen' and undergo an SBT, specific criteria must be met.
  Arms: Once daily screening
Procedure: Twice daily screening — In the 'at least twice daily' screening arm patients will be screened at a minimum between approximately 6:00-8:00 hours and 13:00-15:00 hours daily. To pass the 'readiness to wean screen' and undergo an SBT, specific criteria must be met.
  Arms: At least twice daily screening
Procedure: PS SBTs — Patients are assigned a SBT technique. All SBTs for these patients must be conducted on PS =< 8 cm H2O with PEEP =< 5 cm H2O.
  Arms: PS SBTs
Procedure: T-piece SBTs — Patients are assigned a SBT technique. All SBTs for these patients must be conducted with T-piece.
  Arms: T-piece SBTs

SUMMARY:
The requirement for invasive mechanical ventilation is a defining feature of critical illness. Liberation or weaning is the process during which the work of breathing is transferred from the ventilator back to the patient. Approximately 40% of the time spent on mechanical ventilation is dedicated to weaning. Limiting the duration of invasive ventilation has been identified as a key research priority in critical care. Studies support the use of screening protocols (once daily vs. usual care) to identify weaning candidates and the conduct of tests of patient's ability to breathe spontaneously (SBTs). While once daily screening is the current standard of care in national intensive care units (ICUs), it is poorly aligned with the 24/7 ICU care environment wherein a critically ill patients' status can change from hour to hour. Only one large trial has compared alternative SBT techniques [T-piece vs PS (Pressure Support)]. No trial has compared a strategy of more frequent screening to once daily screening or alternative SBT techniques. The presence of respiratory therapists (RTs) 24/7 in North American ICUs presents a unique opportunity to screen more frequently, conduct more frequent SBTs, and determine the optimal strategy to liberate critically ill adults from invasive ventilation.

The investigators propose to conduct a pilot randomized trial in 100 critically ill adults comparing 'once daily' screening to 'at least twice daily' screening and PS vs. T-piece SBTs in 12 Canadian ICUs. In the proposed trial, the investigators will (i) assess their ability to recruit critically ill adults who can breathe spontaneously or initiate breaths on one of several commonly used modes of ventilation into the trial, (ii) evaluate clinician's ability to implement the trial as designed, (iii) assess current practices in sedation, analgesia and delirium management and timing of patient mobilization prior to conducting screening assessments, (iv) identify barriers (clinician, institutional) to enrolling patients, (v) characterize trial participants based on weaning difficulty, and (vi) obtain preliminary estimates of the impact of the alternative screening and SBT strategies on clinically important outcomes.

DETAILED DESCRIPTION:
Identifying the optimal time when patients are ready to be weaned from invasive ventilation is challenging and often arbitrary. To identify weaning candidates, current guidelines recommend that clinicians use a combination of subjective clinical assessments and objective measurements. However, clinician's subjective assessments of weaning readiness underestimate the probability that patients can be successfully liberated from mechanical ventilation. Even the most objective measurement, the respiratory frequency to tidal volume ratio or rapid shallow breathing index (f/VT), has only limited value [Likelihood ratio + 1.58 (1.30 -1.90)] in predicting successful extubation after a trial of spontaneous breathing trial (SBT).

More than two decades of research support the use of specific strategies to limit the duration of invasive ventilation including the (i) use of multidisciplinary screening protocols to identify SBT candidates, (ii) conduct of SBTs in patients who meet screening criteria, and (iii) use of specific modes and techniques Pressure Support (PS) and once daily SBTs [e.g., PS or T-piece (no support)] to discontinue support in patients who fail an initial SBT and require weaning. Compared to usual care, earlier trials have shown that protocolized weaning, led by allied health care providers (RTs, nurses) reduced weaning time.

A systematic review and meta-analysis of 11 trials involving 1,971 critically ill patients, conducted by one investigative member of the study team (KB), demonstrated that screening protocols reduce the total duration of mechanical ventilation, the time spent weaning and ICU length of stay. Only 1 trial (n=385) compared twice daily screening led by RTs and bedside nurses to usual care (requiring a physician order to conduct an SBT) and found a significantly shorter duration of ventilation and a trend toward a lower ventilator-associated pneumonia (VAP) rate in the twice daily screening group. The investigator's prior work demonstrates that once daily screening is the current standard of care nationally and internationally.

Further, no trial has compared two of the most frequently used SBT techniques internationally [PS and T-piece]. Consequently, little is known about how frequently patients should be screened and what technique should be used to conduct SBTs in Canadian ICUs today. The FAST trial will address these important gaps in knowledge.

The proposed study is novel in seeking to identify the optimal screening and SBT strategies to minimize patients' exposure to invasive ventilation and the complications associated with it. It will evaluate how weaning strategies are delivered to critically ill adults and determine whether alternative delivery strategies may improve patient outcomes. Only one weaning trial has been conducted in Canada previously by members of the investigative team (KB, MM). Establishing the role for more frequent screening is appealing to ICU clinicians (intensivists, RTs, nurses, physiotherapists) because it is a sensible and low-risk intervention that represents a cost-effective use of current resources. Moreover, this simple intervention holds promise as a strategy that could change clinical practice, enhance the care delivered to critically ill adults, and improve patient outcomes.

In the FAST Trial,eligible patients will be randomized to a screening frequency (once vs. at least twice daily) and an SBT technique (PS vs. T-piece). The investigators propose to evaluate the feasibility of conducting an open-label, multicentre, factorial design trial involving 100 critically ill adults which compares screening frequency and SBT technique in 12 Canadian ICUs. In the pilot trial, the investigators will (i) evaluate their ability to recruit the desired population, (ii) assess clinician adherence to the screening and SBT protocols, (iii) identify potential confounders, (iv) characterize trial participants based on weaning difficulty, and (iv) obtain preliminary estimates of the effect of the alternative screening and SBT strategies on important outcomes.

In the pilot trial, the investigative team will also assess 'current practices' with regard to sedation, analgesia, and delirium management, as well as, timing of mobilization prior to screening assessments to identify practices that may bias duration of ventilation and require protocolization in the future, planned large scale weaning trial. All participating adult ICUs currently titrate sedation use to either the Sedation-Agitation Scale (SAS) or Richmond Agitation Sedation Scale (RASS), have dedicated RT personnel present 24 hours per day/7 days per week and have either full time, part time, or consulting Physiotherapists.

The investigators will determine if the proposed multicentre screening randomized control trial (RCT) is:

A. Feasible, specifically, can the investigative team:

1. Recruit critically ill adults breathing spontaneously on Pressure Support (PS) or proportional assist ventilation (PAV), or triggering breaths on volume or pressure Assist Control (AC), volume or pressure Synchronized Intermittent Mandatory Ventilation (SIMV) ± PS, Pressure Regulated Volume Control (PRVC) or Airway Pressure Release Ventilation (APRV) into a trial comparing 'once daily' to 'at least twice daily' screening to identify weaning candidates,
2. Comply with 'once daily' and 'at least twice daily' screening assessment protocols with minimal contamination in 'once daily' arm,
3. Comply with PS and T-piece SBT protocols with minimal contamination in either arm,
4. Quantify potential co-interventions (sedation, analgesia and delirium management and timing of mobilization) that may lead to performance bias and may require protocolization in the future, planned, large scale weaning trial,
5. Identify barriers (clinician and institutional) to recruitment,
6. Classify trial participants as those requiring (i) simple, (ii) difficult or (iii) prolonged weaning using established definitions,
7. Obtain preliminary estimates of the impact of the alternative screening ('once daily' vs. 'at least twice daily') and SBT techniques (PS vs. T-piece) on important outcomes [e.g., time to first SBT and first successful SBT, time to first extubation and successful extubation, total duration of mechanical ventilation, ICU and hospital length of stay, ICU and hospital mortality, the use of noninvasive ventilation (NIV) after extubation

B. Safe, with regard to the proportion of patients experiencing weaning related complications (self-extubation, reintubation, tracheostomy) in both screening and SBT strategies.

Information obtained from the pilot trial will inform the design of the planned large scale trial evaluating the time to first successful SBT completion (SBT outcome) and the time to first successful extubation (weaning and extubation outcome). In this manner, the investigators will assess the feasibility of conducting a multicentre, multinational RCT addressing this important research question.

ELIGIBILITY:
Inclusion Criteria:

The investigators will include patients who are:

1. receiving invasive mechanical ventilation for >= 24 hours.
2. capable of initiating spontaneous breaths on Pressure Support (PS) or Proportional Assist Ventilation (PAV) or triggering breaths on volume or pressure Assist Control (AC), volume or pressure Synchronized Intermittent Mandatory Ventilation (SIMV) ± PS, Pressure Regulated Volume Control (PRVC) or (Airway Pressure Release Ventilation) APRV,
3. with a fraction of inspired oxygen (FiO2) of =< 70% and
4. with a positive end-expiratory pressure (PEEP) of =< 12 cm H2O.

Exclusion Criteria:

The investigators will exclude patients who are

1. admitted after cardiopulmonary arrest or with brain death or expected brain death,
2. who have evidence of myocardial ischemia in the 24 hour period before enrollment,
3. who have received continuous invasive mechanical ventilation for >= 2 weeks,
4. who have a tracheostomy in situ at the time of screening,
5. who are receiving sedative infusions for seizures or alcohol withdrawal,
6. who require escalating doses of sedative agents,
7. who are receiving neuromuscular blockers or who have known quadriplegia, paraplegia or 4 limb weakness or paralysis preventing active mobilization (e.g., active range of motion, exercises in bed, sitting at edge of bed, transferring from bed to chair, standing, marching in place, ambulating),
8. who are moribund (e.g., at imminent risk for death) or who have limitations of treatment (e.g., withdrawal of support, do not reintubate order, however, do not resuscitate orders will be permitted),
9. who have profound neurologic deficits (e.g. large intracranial stroke or bleed) or Glasgow Coma Scale (GCS) < 6,
10. who are using modes that automate SBT conduct,
11. who are current enrolled in a confounding study that includes a weaning protocol, or
12. who were previously enrolled in this trial,
13. patients who have already undergone an SBT or who are on settings compatible with an SBT (T-piece, CPAP without PS (any level), or PS (=< 8 cm H2O regardless of PEEP)
14. patients who have already undergone extubation [planned, unplanned (e.g. self, accidental)] during the same ICU admission.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-07; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Recruitment metrics as measured by number of critically ill patients enrolled per ICU per month | 24 Months
  Assess the investigative team's ability to recruit, on average, 2 invasively ventilated, critically ill adults who can breathe spontaneously or initiate breaths on one of several commonly used modes of ventilation into the trial, per ICU ment per month.

SECONDARY OUTCOMES:
Adherence to protocol as measured by rate of protocol violations | 24 Months
  Evaluate clinician's ability to implement the trial as designed
Current practices regarding sedation, analgesics, delirium and mobilization as assessed using a checklist prior to screening | 24 Months
  Assess current practices in sedation, analgesia and delirium management and timing of patient mobilization prior to conducting screening assessments
Enrollment Barriers as measured by consent rates and presence of exclusion criteria | 24 Months
  Identify barriers (clinician, institutional) to enrolling patients, (v) characterize trial participants based on weaning difficulty
Characterize Weaning as simple, difficult or prolonged according to the Task Force on Weaning definitions | 24 Months
  Characterize trial participants based on weaning difficulty
Clinically Important Outcomes | 24 Months
  Obtain preliminary estimates of the impact of the alternative screening and SBT strategies on clinically important outcomes (i.e. time to first SBT and first successful SBT, time to first extubation and successful extubation, total duration of mechanical ventilation, ICU and hospital length of stay, ICU and hospital mortality, the use of noninvasive ventilation (NIV) after extubation).

CONTACTS AND LOCATIONS:
Overall Officials: Karen Burns, MD, FRCPC, Principal Investigator — St. Michael's Hopsital, Toronto, Canada
Locations (10):
- United States (2):
  - Longbeach Memorial Hospital, Long Beach, California
  - Grady Memorial Hospital, Atlanta, Georgia
- Canada (8):
  - St Paul's Hospital, Vancouver, British Columbia
  - Juravinski Hospital, Hamilton, Ontario
  - St. Joseph's Hospital, Hamilton, Ontario
  - Ottawa Civic Hospital, Ottawa, Ontario
  - Ottawa General Hospital, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - St. Joseph's Hospital, Toronto, Toronto, Ontario
  - Universite de Sherbrooke, Sherbrooke, Quebec

REFERENCES:
- [Derived] Burns KEA, Wong J, Rizvi L, Lafreniere-Roula M, Thorpe K, Devlin JW, Cook DJ, Seely A, Dodek PM, Tanios M, Piraino T, Gouskos A, Kiedrowski KC, Kay P, Mitchell S, Merner GW, Mayette M, D'Aragon F, Lamontagne F, Rochwerg B, Turgeon A, Sia YT, Charbonney E, Aslanian P, Criner GJ, Hyzy RC, Beitler JR, Kassis EB, Kutsogiannis DJ, Meade MO, Liebler J, Iyer-Kumar S, Tsang J, Cirone R, Shanholtz C, Hill NS; Canadian Critical Care Trials Group. Frequency of Screening and Spontaneous Breathing Trial Techniques: A Randomized Clinical Trial. JAMA. 2024 Dec 3;332(21):1808-1821. doi: 10.1001/jama.2024.20631. PMID 39382222
- [Derived] Burns KEA, Lafrienier-Roula M, Hill NS, Cook DJ, Seely AJE, Rochwerg B, Mayette M, D'Aragon F, Devlin JW, Dodek P, Tanios M, Gouskos A, Turgeon AF, Aslanian P, Sia YT, Beitler JR, Hyzy R, Criner GJ, Kassis EB, Tsang JLY, Meade MO, Liebler JM, Wong JTY, Thorpe KE; Canadian Critical Care Trials Group. Frequency of screening and SBT Technique Trial-North American Weaning Collaboration (FAST-NAWC): an update to the protocol and statistical analysis plan. Trials. 2023 Oct 2;24(1):626. doi: 10.1186/s13063-023-07079-5. PMID 37784109
- [Derived] Burns KEA, Rizvi L, Cook DJ, Seely AJE, Rochwerg B, Lamontagne F, Devlin JW, Dodek P, Mayette M, Tanios M, Gouskos A, Kay P, Mitchell S, Kiedrowski KC, Hill NS; Canadian Critical Care Trials Group. Frequency of Screening and SBT Technique Trial - North American Weaning Collaboration (FAST-NAWC): a protocol for a multicenter, factorial randomized trial. Trials. 2019 Oct 11;20(1):587. doi: 10.1186/s13063-019-3641-8. PMID 31604480